CLINICAL TRIAL: NCT01726569
Title: A Randomized Trial of the Impact of Multifaceted Education on Post-operative Satisfaction With Glaucoma Surgery in Rural China
Brief Title: Post-operative Satisfaction With Glaucoma Surgery Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study sites were reconsidered.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Congdon Nathan, Guangdong Educational Intervention for Rural Glaucoma surgical patient, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ZOC-CREST1
Record Dates: First submitted 2012-11-10; First posted 2012-11-15 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Glaucoma
Keywords: glaucoma; educational intervention; post-operative satisfaction; knowledges
MeSH Terms: conditions — Glaucoma | interventions — Motion Pictures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- film and trained counseling (Experimental): Subjects will be asked to watch a 5-10 min film and participate in a 10-15 min pre-operative counseling session with a trained doctor/nurse. Subjects will also participate in a 5 min post-operative counseling session and follow up counseling after operation 1 week and 6 weeks
  Interventions: Behavioral: film and trained counseling; Other: traditional counseling
- traditional counseling (Other): Subjects will be participate or not participate in pre-operative counseling and/or post-operative counseling with a rural hospital's doctor/nurse.
  Interventions: Other: traditional counseling

INTERVENTIONS:
Behavioral: film and trained counseling — Subjects will be asked to watch a 5-10 min film and participate in a 10-15 min pre-operative counseling session with a trained doctor/nurse. Subjects will also participate in a 5 min post-operative counseling session.
  Arms: film and trained counseling
Other: traditional counseling — Subjects will be not participate or participate in a pre-operative/post-operative counseling session with a rural hospital's doctor/nurse as usual traditional methods.

SUMMARY:
1. Investigate degree of postoperative satisfaction in county level hospital glaucoma patients.
2. Investigate the effect of educational intervention affect the degree of satisfaction in glaucoma patients.
3. Investigate the effect factors of postoperative satisfaction.

DETAILED DESCRIPTION:
Glaucoma is the leading cause irreversible blindness worldwide, but only less than 10% glaucoma patients were diagnosed in the country of Asia areas. In the country of China, patients who are low educational level and less known acknowledgement and information have less known glaucoma. In the help of the government and some international non-governmental organizations(NGOs), a lot of people in the country know the cataract, and the operability of cataract is increase. Because vision loss usually development after operation for glaucoma. If patients did not understand this, they may be not only do not accept operation, but also affect operability of cataract. We hope the educational intervention for glaucoma can increase the degree of satisfaction in glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years, glaucoma patients who do the peripheral iridectomy or trabeculotomy

Exclusion Criteria:

* patients who had been the trabeculotomy, vision≤0.05, severe psychotic disorders and dysgnosia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
postoperative satisfaction rate in both group | after surgery up to 6 weeks
  the rate of satisfaction

SECONDARY OUTCOMES:
knowledge about glaucoma | before surgery and after surgey 1 week and 6 weeks
  the knowledge about glaucoma scores
willingness to recommend surgery | after surgery 1 week and 6 weeks
  The rate of willingness to recommend surgery
personality in both groups | Baseline (before surgery)
  use Eysenck Personality Questionnaire-Revised Short Scale for Chinese(EPQ_RSC) access glaucoma patients personality
intraocular pressure and visual acuity in both groups | before surgery and after surgery 1week and 6 weeks
  intraocular pressure and visual acuity in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Congdon, MD,MPH, Principal Investigator — Zhongshan Ophthalmic Center,Sun Yat-sen University;ORBIS
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China